CLINICAL TRIAL: NCT02108405
Title: The Value of Memory B Cells Marker (CD27) and Howell Jelly Bodies Detrection in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant professor, Tanta University
Other Study IDs: 1020/02/13
Record Dates: First submitted 2013-03-01; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Sepsis
Keywords: critically ill patient.
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis: Sepsis Forty eight patients developed septic complication during ICU stay (sepsis group).
- SIRS group: SIRS group Forty seven patients were critically ill without evidence of infectious organism (SIRS group).

SUMMARY:
A total of ninety - five patients (54men and 41women) were included in the study. Fifty-eight patients developed septic complication during ICU stay (sepsis group). Forty seven patients were critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis were measured. Routine cultures were obtained. The attending physician evaluated the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. Memory B cells and Heinz bodies were monitored.

DETAILED DESCRIPTION:
The patients staying in ICU for more than 24 hours were enrolled in the study. Patients received anti-inflammatory drugs or corticosteroids before admission, patients had immunosuppressive illness, patients had chronic organ failure; patients received massive blood transfusion; patients with radiation therapy and patients with previous organ transplantation were excluded from the study. At admission, patient's age, sex, weight and height were recorded. Patients data that include the clinical status; sequential organ failure assessment (SOFA) score; temperature; heart rate; respiratory rate; blood pressure; central venous pressure; laboratory analysis (complete blood count, blood urea nitrogen, blood sugar, serum sodium, potassium, calcium, aspartate aminotransferase, alanine aminotransferase, prothrombin time, albumin and CRP) and arterial blood gas analysis were measured. Routine cultures of suspected sites, blood and urine were obtained to determine the presence of infection. We attempted to maintain the patient hemoglobin level at 10-12g/dl and central venous pressure at 8-12 cmH2o. When needed, intravascular fluid replacement, blood products and inotropic or vasopressor agents were administered. Each day the attending physician evaluated all the study patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with manifestation of sepsis or SIRS

Exclusion Criteria:

* Patients received anti-inflammatory drugs or corticosteroids before admission, who had immunosuppressive illness, who had chronic organ failure; who had received massive blood transfusion; those with radiation therapy, previous organ transplantation were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of ninety five patients were included in the study. fifty eight patients developed septic complication during ICU stay (sepsis group). fifty seven patients were critically ill without evidence of infectious organism (SIRS group). At admission, the patient's age, sex, height and weight were recorded.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Memory B cells | 1 day (At time of ICU admission)
  Memory B cells detection was made using flowcytometry.

SECONDARY OUTCOMES:
Heinz bodies | 1 day (At ICU admission)
  Heinz bodies using flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant Professor
Locations (1):
- Tanta University, Tanta, Algharbyia, Egypt